CLINICAL TRIAL: NCT04698915
Title: GRECO-2: A Randomized, Phase 2b Study of GC4711 in Combination With Stereotactic Body Radiation Therapy (SBRT) in the Treatment of Unresectable or Borderline Resectable Nonmetastatic Pancreatic Cancer
Brief Title: Phase 2b Study of GC4711 in Combination With SBRT for Nonmetastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility Analysis
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTI-4711-201
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: SBRT; Borderline Resectable Pancreatic Cancer; Unresectable Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A Active GC4711 (Experimental)
  Interventions: Drug: Drug GC4711
- Arm B Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug GC4711 — 15 Minute IV Infusion
  Arms: Arm A Active GC4711
Drug: Placebo — 15 Minute IV Infusion
  Arms: Arm B Placebo

SUMMARY:
GTI-4711-201 is designed as a Phase 2b, multicenter, randomized, double-blind, placebo-controlled study to determine the effect to OS by adding GC4711 to SBRT following chemotherapy in patients with unresectable or borderline resectable nonmetastatic

ELIGIBILITY:
Inclusion Criteria:

1. Histological or biopsy proven adenocarcinoma of the pancreas. Cytology is acceptable if histology cannot be obtained.
2. Newly diagnosed non-metastatic PC judged by tumor board to be feasible for SBRT
3. Completed at least 6 weeks of chemotherapy consisting of FOLFIRINOX, mFOLFIRINOX, or a gemcitabine-based doublet regimen prior to start of SBRT
4. Remain non-metastatic as confirmed by a CT scan at screening.
5. Female or male subjects ≥ 18 years of age
6. ECOG performance status of 0-2
7. Adequate end-organ function

Exclusion Criteria:

1. Subjects with documented metastatic disease
2. First-line chemotherapy other than FOLFIRINOX, mFOLFIRINOX, and/or a gemcitabine-based doublet regimen
3. Prior abdominal RT with substantial overlap in radiation fields
4. Subjects not recovered/controlled from treatment-related toxicities
5. Uncontrolled malignancy other than PC
6. Uncontrolled gastric or duodenal ulcer disease within 30 days of dosing
7. Visible invasion of bulky tumor into the lumen of the bowel or stomach on endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (21):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Miami, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Northwell Health, Lake Success, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Radiation Oncology and Gamma Knife Center of Oregon, Portland, Oregon
  - Pennsylvania State University, University Park, Pennsylvania
  - UT Southwestern Medical, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center (UWMC) - Radiation Oncology Center, Seattle, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
- Canada (3):
  - London Regional Cancer Center, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Atlantic Clinical Cancer Research Unit/QEII Health Sciences Centre, Halifax, Nova Scotia
- France (6):
  - Institut Bergonié, Bordeaux
  - CHRU de Brest Hôpital Morvan, Brest
  - Centre Georges François Leclerc, Dijon
  - Institut régional du Cancer de Montpellier, Montpellier
  - Tenon Hospital, Paris
  - CHU de Bordeaux, Hôpital Haut-Lévêque, Pessac
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeenshire
  - GenesisCare, Oxford, Oxfordshire
  - Addenbrookes Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Imperial College London, Saint Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffe SE, Aguilera TA, Parikh PJ, Ghaly MM, Herman JM, Caster JM, Kim DW, Costello J, Malafa MP, Moser EC, Kennedy EP, Terry K, Kurman M. Stereotactic body radiotherapy plus rucosopasem in locally advanced or borderline resectable pancreatic cancer: GRECO-2 phase II study design. Future Oncol. 2024 Mar;20(8):437-446. doi: 10.2217/fon-2022-1219. Epub 2024 Jan 24. PMID 38264869
- [Derived] Taniguchi CM, Frakes JM, Aguilera TA, Palta M, Czito B, Bhutani MS, Colbert LE, Abi Jaoude J, Bernard V, Pant S, Tzeng CD, Kim DW, Malafa M, Costello J, Mathew G, Rebueno N, Koay EJ, Das P, Ludmir EB, Katz MHG, Wolff RA, Beddar S, Sawakuchi GO, Moningi S, Slack Tidwell RS, Yuan Y, Thall PF, Beardsley RA, Holmlund J, Herman JM, Hoffe SE. Stereotactic body radiotherapy with or without selective dismutase mimetic in pancreatic adenocarcinoma: an adaptive, randomised, double-blind, placebo-controlled, phase 1b/2 trial. Lancet Oncol. 2023 Dec;24(12):1387-1398. doi: 10.1016/S1470-2045(23)00478-3. PMID 38039992
- [Derived] Squillace S, Salvemini D. Nitroxidative stress in pain and opioid-induced adverse effects: therapeutic opportunities. Pain. 2022 Feb 1;163(2):205-213. doi: 10.1097/j.pain.0000000000002347. No abstract available. PMID 34145168

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A Active GC4711 | Arm B Placebo
Started | 84 | 84
Completed | 0 | 0
Not Completed | 84 | 84
Not completed — Adverse Event | 2 | 0
Not completed — Death | 23 | 20
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study Terminated by Sponsor | 55 | 60
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat Population that includes all randomized subjects that received at least one dose of GC4711/Placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Active GC4711 | Arm B Placebo | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 38 | 74
  >=65 years | 48 | 46 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 86
  Male | 40 | 42 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 70 | 67 | 137
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to the date of death from any cause. The number of subjects that have died during this time period is the reported outcome measure.
Time Frame: From randomization of the first subject until 30 days post last dose of GC4711/ and SBRT for the last subject randomized to the study (total duration 2years and 6.5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Active GC4711 | Arm B Placebo
Number analyzed (Participants) | 84 | 84
Participants | 24 | 20

ADVERSE EVENTS:
Time Frame: All AEs/SAES were monitored/assessed from time of randomization until up to 30 days post the last dose of GC4711/Placebo (2 months). Since the primary endpoint of the trial was overall survival, deaths were assessed for a longer duration than AEs/SAEs. Due to the study being terminated early, all subject death information was collected for a minimum of 30 days post the last dose of GC4711/Placebo (2months)
Arm/Group | Arm A Active GC4711 | Arm B Placebo
All-Cause Mortality (participants affected / at risk) | 24/84 | 20/84
Serious Adverse Events (participants affected / at risk) | 17/84 | 14/84
Other Adverse Events (participants affected / at risk) | 76/84 | 71/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Active GC4711 (N=84) | Arm B Placebo (N=84)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fistula of Small Intestine (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalised Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 0 (0)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Cholecystitis Infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colititis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Peripancreatic fluid Collection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 2 (2) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Device Occlusion (Product Issues) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphatic Fistula (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Active GC4711 (N=84) | Arm B Placebo (N=84)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 8 (8)
Abdominal Distension (Gastrointestinal disorders) | 7 (7) | 8 (8)
Abdominal Pain (Gastrointestinal disorders) | 16 (16) | 16 (16)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 13 (13)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 44 (44) | 32 (32)
Vomiting (Gastrointestinal disorders) | 26 (26) | 15 (15)
Fatigue (General disorders) | 38 (38) | 26 (26)
Alanine aminotransferase increased (Investigations) | 5 (5) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 10 (10) | 4 (4)
Blood Bilirubin Increased (Investigations) | 5 | 1
Lymphocyte count decreased (Investigations) | 8 (8) | 3 (3)
Platelet Count Decreased (Investigations) | 4 (4) | 6 (6)
White Blood Cell Count Decreased (Investigations) | 5 (5) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9)
Dizziness (Nervous system disorders) | 15 (15) | 6 (6)
Headache (Nervous system disorders) | 8 (8) | 4 (4)
Paraesthesia (Nervous system disorders) | 8 (8) | 4 (4)
Insomnia (Psychiatric disorders) | 5 (5) | 2 (2)
Hypertension (Vascular disorders) | 8 (8) | 10 (10)
Hypotension (Vascular disorders) | 18 (18) | 3 (3)

LIMITATIONS AND CAVEATS:
Study was terminated early by the Sponsor based on a futility analysis that was conducted in which the trial met the prespecified early termination rules. The last randomized subject did not complete protocol therapy but was followed for safety for a period of 30 days post the last administration of GC4711/Placebo +SBRT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04698915/Prot_SAP_000.pdf